CLINICAL TRIAL: NCT01641887
Title: Personalized Decision Aid for the Management of Gastroesophageal Reflux Disease
Brief Title: Decision Aid for Gastroesophageal Reflux Disease Management
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Chin Hur, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2012-MGH-Hur-GERD
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Gastroesophageal Reflux Disease; Esophageal Cancer; Barrett's Esophagus
Keywords: GERD; Heartburn; Decision Aid
MeSH Terms: conditions — Gastroesophageal Reflux; Esophageal Neoplasms; Barrett Esophagus; Heartburn | interventions — Decision Support Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GERD patients: Patients who have GERD will be recruited for this study.
  Interventions: Other: Decision Aid

INTERVENTIONS:
Other: Decision Aid — Patients will use a decision aid administered on a computer.

SUMMARY:
The study is to test a decision aid that is designed to help patients make decision regarding management of their gastroesophageal reflux disease (GERD). Once the decision aid is constructed we will test and assess the aid on ~100 patients who have GERD to assess effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GERD,
* Age at least 18,
* Able to give consent

Exclusion Criteria:

* Unable to perform decision aid on a computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have GERD who have not yet had endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Participant acceptability | Patients will be surveyed on the day of the decision aid (1 day).
  Patients will be surveyed after using the intervention to determine if they felt it was useful and whether they would recommend it to others.
Participant Satisfaction | Patients will be surveyed on the day of the decision aid (1 day).
  The Patient Satisfaction with Decision Scale will be adapted for this study. This is a six-item scale has been shown to be reliable and valid.

SECONDARY OUTCOMES:
Patient decisions | Patients will be surveyed on the day of the decision aid (1 day).
  Patient intervention choice will be solicited both before and after the decision aid.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States